CLINICAL TRIAL: NCT03136770
Title: A Randomized, Open-label, Two-way Crossover Study to Assess the Pharmacokinetics and Safety of CK-30 600 mg (Compound K) and Red Ginseng Extracts 2.94 g After a Single Oral Dose in Healthy Male Volunteers
Brief Title: A Randomized, Open-label, Two-way Crossover Study to Assess the Pharmacokinetics and Safety of CK-30 600 mg (Compound K)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In-Jin Jang, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CK-30
Record Dates: First submitted 2017-01-31; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): CK-30 600 mg -> red ginseng extracts 2.94 g
  Interventions: Dietary Supplement: CK-30; Dietary Supplement: Red ginseng extracts
- B (Experimental): red ginseng extracts 2.94 g -> CK-30 600 mg
  Interventions: Dietary Supplement: CK-30; Dietary Supplement: Red ginseng extracts

INTERVENTIONS:
Dietary Supplement: CK-30 — Compound K 600 mg
Dietary Supplement: Red ginseng extracts — Red ginseng extracts 2.94 g

SUMMARY:
A study to assess the pharmacokinetics and safety of CK-30 600 mg (Compound K) and red ginseng extracts 2.94 g after a single oral dose in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Koreans between 19 and 45 years of age at the screening
* A body weight of greater than 55 kg, and a body mass index (BMI) of between 18.0 and 27.0, wherein BMI (kg/m2) = Weight (kg) / [Height (m)]2
* Full understanding of all the information regarding this clinical trial after listening to a detailed explanation, deciding to participate in the clinical trial by one's own will, and signing a written consent to comply with the precautions

Exclusion Criteria:

* History of herbal medicine including ginseng and red ginseng extracts within 2 weeks before the first administration of the IP
* Present condition or history of any clinically significant disease in the liver, nervous system, immune system, respiratory system, or endocrine system; hematologic or oncologic disease; cardiovascular disease; or psychiatric disorder (mood disorder, obsessive-compulsive disorder, etc.)
* Clinical evidence or history of gastrointestinal disease (including Crohn's disease, gastric ulcer, and acute or chronic pancreatitis) or history of gastrointestinal surgery (except for appendectomy or hernia surgery) that could affect the pharmacokinetic and safety assessment of the IP
* Clinical evidence of genetic disorders such as galactose intolerance, Lapp lactose deficiency, and/or glucose-galactose malabsorption
* History of hypersensitivity, including drug allergy (red ginseng extracts, aspirin, antibiotics, etc.), or history of clinically significant hypersensitivity
* Meeting the following criteria at the screening: Serum AST (SGOT) or ALT (SGPT) > 1.5 times the upper normal limit
* History of drug abuse, or a positive reaction to an abusive drug in a urine drug screening
* Having taken any prescribed medicine or herbal supplement within two weeks before the first administration of the IP, or any non-prescribed medicine or vitamin supplement within one week before the first administration of the IP (If the other conditions were satisfied, the subject could be deemed eligible for the trial at the discretion of the investigator.)
* Participation in and administration of the IP of another clinical trial within three months before the first administration of the IP
* Donation of a unit of blood within two months, or of blood components within one month, or receipt of a blood transfusion within one month before the first administration of the IP
* Consumption of more than 21 units of alcohol per week (one unit being 10 g of pure alcohol) or inability to abstain from drinking alcohol during the study period
* History of smoking 10 cigarettes per day within three months before the first administration of the IP (Subjects who quit smoking for at least three months before the first administration of the IP can still be enrolled in the trial.) or subjects who are not able to quit smoking from 24 hours before hospitalization to discharge.
* Consumption of grapefruit-containing products within 24 hours before the hospitalization or inability to abstain from consuming grapefruit-containing products during the study period
* Subjects who are not able to abstain from drinking caffeine-containing products (coffee, tea), carbonated drinks, nutrient tonics during the study period
* For females, plan to conceive or become pregnant, or inability to use an appropriate method of contraception (e.g., sterilization operation of the subject or his partner, intrauterine device of the partner, a barrier contraceptive method, or a combination of the diaphragm and condom methods) during the study period
* Assessment as ineligible by the investigator based on the results of the clinical laboratory tests or other assessments

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax) | Total 16 days
  Pharmacokinetics of CK-30 and Red ginseng extracts
Pharmacokinetics (AUClast) | Total 16 days
  Pharmacokinetics of CK-30 and Red ginseng extracts

SECONDARY OUTCOMES:
Safety and tolerability (Number of participants with treatment-related adverse events) | Total 16 days
  Safety of CK-30 and Red ginseng extracts

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital Clinical Trials Center, Seoul, South Korea

REFERENCES:
- [Result] Jin H, Seo JH, Uhm YK, Jung CY, Lee SK, Yim SV. Pharmacokinetic comparison of ginsenoside metabolite IH-901 from fermented and non-fermented ginseng in healthy Korean volunteers. J Ethnopharmacol. 2012 Jan 31;139(2):664-7. doi: 10.1016/j.jep.2011.11.052. Epub 2011 Dec 9. PMID 22178175
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed?term=Pharmacokinetic+comparison+of+ginsenoside+metabolite+IH-901+from+fermented+and+non-fermented+ginseng+in+healthy+Korean+volunteers&TransSchema=title&cmd=detailssearch